CLINICAL TRIAL: NCT02165878
Title: KoreaN Cohort Study for Outcome in Pediatric Patients With Chronic Kidney Disease : A 10-year Longitudinal Cohort Study of the Chronic Kidney Disease
Brief Title: KoreaN Cohort Study for Outcome in Pediatric Patients With Chronic Kidney Disease
Acronym: KNOW-PedCKD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Jeju National University Hospital (Other); Pusan National University Hospital (Other); Samsung Medical Center (Other); Kyungpook National University Hospital (Other); Yonsei University (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Il Soo Ha, Professor, Seoul National University Hospital
Other Study IDs: 2013E3301601; KNOW-PedCKD (Other: Seoul National University Hospital)
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: Chronic kidney disease(CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A biobank is also established for the DNA, serum and urine taken at regular interval.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children and adolescent: children and adolescent CKD patients of any etiology

SUMMARY:
KNOW-CKD (KoreaN cohort study for Outcome in patients With Chronic Kidney Disease) is a nation-wide, ten-year longitudinal cohort study, launched in 2011. The aim of the study is to assess the characteristics and risk factors of progression and complications of CKD of Korea. Pediatric sub-cohort of KNOW-CKD is planned to enroll 450 children with CKD, stage I to V (pre-dialysis).

DETAILED DESCRIPTION:
Seven major pediatric nephrology centers of Korea enrolled children younger than 20 years who had CKD. Medical history taking, questionaire assessment of socio-economic status, anthropometric measurement, and clinical assessment using laboratory and imaging tests were done. Outcome is development of LV hypertrophy or hypertension, growth, neuropsychological status, behavioral status, kidney growth, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age: < 20 yr
* CKD stage 1 through 5 of KDIGO guideline
* predialysis

Exclusion Criteria:

- Dialysis

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: CKD stage 1 through 5 Ages below 20
Sampling Method: Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
eGFR | 10 years
  eGFR in mL/min/1.73 m2

SECONDARY OUTCOMES:
Development of cardiovascular disease | 10 years
  Hypertrophy in g/m2
Metabolic bone disease | 10 years
  Bone Dexametry in z score
Anemia | 10 years
  Anemia in g/dL
Growth | 10 years
  Height in z score
Health-related quality of life (HRQOL) | 10 years
  PedsQL 4.0 Generic Core Scale Module (Mapi Research Trust, on behalf of Dr James W. Varni, copyright owner of PedsQL™)
Cognitive skills and emotional development | 10 years
  K-WAIS score

CONTACTS AND LOCATIONS:
Overall Officials: Il Soo Ha, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang NR, Ahn YH, Park E, Lee KH, Baek HS, Kim SH, Cho H, Cho MH, Shin JI, Lee JH, Cheong HI, Kang HG, Park YS, Ha IS, Moon DS, Han KH. Intellectual Functioning of Pediatric Patients with Chronic Kidney Disease: Results from the KNOW-Ped CKD. J Korean Med Sci. 2021 May 24;36(20):e138. doi: 10.3346/jkms.2021.36.e138. PMID 34032031
- [Derived] Baek HS, Kim SH, Kang HG, Choi HJ, Cheong HI, Ha IS, Han KH, Cho HY, Shin JI, Park YS, Lee JH, Ahn YH, Park E, Cho MH. Dyslipidemia in pediatric CKD patients: results from KNOW-PedCKD (KoreaN cohort study for Outcomes in patients With Pediatric CKD). Pediatr Nephrol. 2020 Aug;35(8):1455-1461. doi: 10.1007/s00467-020-04545-z. Epub 2020 Mar 30. PMID 32232640
- [Derived] Kang NR, Ahn YH, Park E, Choi HJ, Kim SH, Cho H, Cho MH, Shin JI, Lee JH, Park YS, Cheong HI, Kang HG, Ha IS, Kwack YS, Han KH. Mental health and psychosocial adjustment in pediatric chronic kidney disease derived from the KNOW-Ped CKD study. Pediatr Nephrol. 2019 Oct;34(10):1753-1764. doi: 10.1007/s00467-019-04292-w. Epub 2019 Jun 20. PMID 31222663
- [Derived] Kang HG, Choi HJ, Han KH, Kim SH, Cho HY, Cho MH, Shin JI, Lee JH, Lee J, Oh KH, Park YS, Cheong HI, Ahn C, Ha IS. KNOW-Ped CKD (KoreaN cohort study for outcomes in patients with pediatric CKD): Design and methods. BMC Nephrol. 2016 Mar 25;17:35. doi: 10.1186/s12882-016-0248-0. PMID 27012243